CLINICAL TRIAL: NCT03046329
Title: Improving the Quality of Multiple Myeloma Treatment With Patient Care Plans: Pilot Testing the Impact of Continuing Education and Care Planning on Symptom Management
Brief Title: Improving the Quality of Multiple Myeloma Treatment With Patient Care Plans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carevive Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: G401
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: patient care planning
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Carevive CPS — This intervention will focus on the use of the Carevive CPS at the point of care to enable providers to deliver evidence-based and personalized supportive care and symptom management plans to their MM patients receiving active treatment. The Carevive CPS collects electronic patient reported outcomes (ePROs) and clinical data, reported and entered by clinical staff and/or extracted from the electronic medical record (EMR), and uses these to auto-generate the personalized care plans. Care plan content is driven by practice guidelines and other peer-reviewed evidence, and includes patient education, resources, and referrals developed by expert cancer clinicians and researchers.

SUMMARY:
The overarching objective of this study is to evaluate the symptom assessment and management behaviors used by multiple myeloma (MM) providers for alignment with evidence-based practices, and to explore changes in these symptom care behaviors from baseline to following use of the Carevive Care Planning System (CPS). The overarching goal of the larger program of research is to evaluate the impact of the platform on symptom assessment and management strategies with individuals receiving treatment for multiple myeloma. The current study is focused on determining feasibility of research methods and effect size finding so as to gather the requisite data needed to design fully powered hypothesis testing studies.

DETAILED DESCRIPTION:
Treatment of multiple myeloma (MM) is currently undergoing rapid transformation. With so many new agents and regimens to choose from, significant practice gaps have emerged in the treatment and management of newly diagnosed MM patients. Innovative strategies are needed to (1) enhance the personalized treatment of MM and (2) proactively identify, assess, and manage disease- and treatment-related symptoms so that new therapies are optimally translated to practice. This study will explore the symptom assessment and management practices of providers caring for individuals receiving active therapy for multiple myeloma, and will also employ a two-part intervention (with both patients and providers) to evaluate the impact of a novel existing technology, the Carevive Care Planning System (CPS), on supportive care and symptom management for multiple myeloma patients. The primary objective of this study is to evaluate provider adherence to evidence-based practices for symptom assessment and management (i.e., "symptom care behaviors") of physicians and nurses (providers) caring for individuals receiving active treatment for multiple myeloma (MM). Carevive. The Carevive intervention will include personalized supportive care and symptom management plans for patients auto-generated by the Carevive CPS based on each individual's data. The Care plans were created based on nationally recognized National Comprehensive Cancer Network (NCCN) supportive care guidelines and validated by a Multiple Myeloma (MM) nurse and physician experts. Investigators will use a study-specific scorecard of evidence-based symptom assessment and management metrics to evaluate adherence of provider (n=8-20) symptom assessment and management behaviors, measured at the individual patient (n=120) level, to evidence-based practices for symptom care. Changes in adherence to evidence-based practices will be explored using an across subject comparison to retrospective data abstracted from a matched sample of historical controls. Use of a care planning technology to provide tailored education and individualized information may provide an easy, accessible and effective way to improve supportive care and symptom management for individuals receiving active treatment for multiple myeloma.

Multiple myeloma (MM) is a neoplastic plasma-cell disorder characterized by clonal proliferation of malignant plasma cells in the bone marrow microenvironment, monoclonal protein in the blood or urine, and associated organ dysfunction. In 2014, approximately 24,050 new cases of MM will be diagnosed and 11,090 deaths are expected to occur. The treatment of MM is currently undergoing a rapid evolution. The FDA has approved several new agents over the past several years. Dozens of regimens are now available, with best practices and consensus guidelines continually evolving as new data are published. Indeed, major updates to the International Myeloma Working Group (IMWG) and the 2014 National Comprehensive Cancer Network (NCCN) guidelines highlight the recent revolution in MM care.

With so many agents and regimens to choose from, it is more crucial now than ever for providers to understand how to individualize treatment and symptom management based on patient- and disease-related factors. However, significant practice gaps exist among providers treating patients newly diagnosed with MM. Transplant eligibility, cytogenetics, comorbidities, renal function, and other factors are often not adequately considered when designing personalized induction, consolidation, and maintenance treatment plans. In addition, institutional MM pathways often do not include symptom management. Adverse events are common in patients with MM, and can be dose limiting, forcing patients to change therapies and jeopardize treatment outcomes.

A between subject design using matched historical controls from each institution will be used to evaluate adherence of provider (n=8-20) symptom assessment and management behaviors, measured at the individual multiple myeloma (MM) patient (n=120) level, to evidence-based practices for symptom care, and to explore correlates of adherence to these evidence-based symptom care behaviors. Retrospective reviews of enrolled patient participant charts will be conducted to evaluate achievement of adherence to evidence-based practices at the individual patient level, following engagement with the two part study intervention, plus a novel individualized care planning technology (Carevive CPS). Retrospective chart reviews will be completed on de-identified, matched historical controls (matching on demographics, diagnosis and treatment variables) at each institution (e.g Cleveland Clinic) to assess the impact of the project intervention on the outcome metrics. Data will be entered into the score card appendix B. The use of matched historical controls for comparative analyses addresses the threat of diffusion of intervention; i.e., that participation in this project will have an impact on provider's clinical behaviors in caring for all patients and thus would potentially effect baseline data collection on patients enrolled later on in the study. Providers will be caring for individuals receiving active treatment for multiple myeloma (MM).

The Carevive CPS intervention will focus on the use of the Carevive CPS at the point of care to enable providers to deliver evidence-based and personalized supportive care and symptom management plans to their MM patients receiving active treatment. The Carevive CPS collects electronic patient reported outcomes (ePROs) and clinical data, reported and entered by clinical staff and/or extracted from the electronic medical record (EMR), and uses these to auto-generate the personalized care plans. Care plan content is driven by practice guidelines and other peer-reviewed evidence, and includes patient education, resources, and referrals developed by expert cancer clinicians and researchers. Changes in symptom assessment and management behaviors will be assessed by matching against a scorecard of evidence-based symptom assessment and management metrics. A scorecard metric is being developed by an interdisciplinary team and will be informed by similar approaches used within the Oncology Nursing Society's (ONS) Quality Initiative. Recommendations for symptom assessment and management as well as other evidence based recommendations will be operationalized as metrics.

The intervention is centered on use of the Carevive CPS at the point of care, in conjunction with two consecutive clinical visits, baseline and the second, similar questionnaire will be completed at a clinic visit that occurs at least 4 weeks later. Eligible patients and potentially eligible visits will be identified via weekly chart review of upcoming clinic schedules and of corresponding individual patient medical records. In the exam room, prior to their potential baseline study visit, the patient will be approached and informed of the study (for follow-up visits, patients will be approached and reminded of the study). Once a patient has consented, research staff will open the electronic questionnaire via the Carevive CPS application on one of the study designated tablet computers or secure Cleveland Clinic desktop device according to patient preference . Research staff will then either a) register the patient using their year of birth and a unique Study ID numbers assigned by the Cleveland Clinic or b) open the patients' already existing file (follow-up). The research staff will then select and open the appropriate questionnaire (baseline or interim) and allow the patient to complete. The patient will report their symptoms, history, and current concerns. Once the patient has completed the questionnaire, the survey window will automatically close. Data will be stored centrally and managed by a third party (PRS) in a HIPAA compliant manner. The study research coordinator will then enter limited clinical data into the Diagnosis and Treatment Summary section of the Carevive CPS and click submit. Once submitted, the total composite of ePRO and research staff entered data will run through the guideline-driven and proprietary Carevive CPS algorithms to auto-generate a draft supportive care plan. The draft care plan contains, based on individual patient data, personalized supportive care and symptom management data to be reviewed by the provider during visit. The patient will proceed to the intervention visit where the provider will review, edit if needed, finalize and deliver the electronic care plan (and/or a print copy) to each patient. The patient will also be provided with his or her own copy of the care plan (electronically via email, thumb drive and/or paper) to take home.

Research staff will track patient enrollment and monitor return visits for all participants that fall within the follow-up visit window which begins at least 4 weeks later (+/- 1 week) and continues until the second survey is completed. At this follow up visit, the study patients will take their second electronic survey in the Carevive CPS, and receive their second provider-approved care plan. Patients will also be offered the opportunity to complete a brief questionnaire on their satisfaction with, and utilization of, the care plan since their first intervention visit. The questionnaire will ask about specific recommendations made within the care plan and if the patient recalls receiving it and what action, if any, they have taken. Patients will be offered the opportunity to complete this survey on the study provided tablet or secure Cleveland Clinic desktop device at the time of their second visit or to have a link to the survey emailed to them to be completed at their leisure. This survey will be completed independently of the Carevive CPS through the on-line survey hosting site Surveymonkey.com and will be optional for patients.

Study-specific data collection will occur at multiple time points. Chart reviews of enrolled patient participants will the period of time from baseline intervention (baseline visit) to 12-weeks post the second intervention (encompassing the follow-up visit). Retrospective chart abstractions for the matched controls examine a 12-week time period matched as close as possible to the intervention time period of their respective enrolled patients. Retrospective chart reviews can occur at any time. Chart reviews must reflect the time period of enrolled patients. Patient satisfaction and utilization questionnaire will be completed at or following the follow-up visits. Data sources include the patient questionnaire, previously collected data collected as part of the study intervention and stored within the Carevive CPS platform database (for enrolled patients) limited diagnosis and treatment data on controls (for matching purposes), as well as chart review score card data. A brief worksheet collecting care plan delivery variables (e.g., who delivered the care plan to the patient, how much time was spent reviewing the care plan, etc.) will also be completed by the research staff following each clinic visit at which a care plan is delivered.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Diagnosed with MM and currently receiving treatment
* Receiving active treatment for at least 4 weeks prior to study enrollment

Exclusion Criteria:

* Any participant who cannot understand written or spoken English
* Any participant who is not competent to provide informed consent
* Any participant who cannot be present for the related study visits and/or complete the post-test assessment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Level of provider adherence to evidence-based practices for symptom assessment/management according to chart abstractions | Year 1
  Charts will be abstracted and data will be entered into scorecards to determine whether participating providers adhered to evidence-based practices for symptom assessment and management for study participants.
Degree of changes in symptom care behaviors following engagement with the supportive care intervention according to chart abstractions | Year 1
  Charts will be abstracted and data will be entered into scorecards to explore changes in symptom care behaviors following engagement with a supportive care intervention (the Carevive CPS), and compare to adherence rates for historical controls from the pre-intervention period.

SECONDARY OUTCOMES:
Time spent delivering care plans at both baseline and follow-up using self-report by clinicians | Year 1
  Clinicians will complete a qualitative survey at the end of the study to report the amount of time they spent reviewing and delivering care plans with study participants.
Level of patient satisfaction and utilization of care plans using the SUS survey | Year 1
  The study will explore patient satisfaction and utilization of care plans by asking patients a series of qualitative questions.

IPD SHARING:
Plan to Share IPD: No